CLINICAL TRIAL: NCT04551144
Title: Effect of Transgender Therapy on Hormone Receptors, Adipogenesis, Myogenesis and Inflammation
Brief Title: Effect of Transgender Therapy on Muscle, Fat and Tissue Receptors
Status: Terminated | Type: Observational
Why Stopped: lack of recruitment
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Sandeep Singh Dhindsa, M.D., F.A.C.E, Professor of Medicine, St. Louis University
Other Study IDs: 31184
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Gender Incongruence; Transgenderism
MeSH Terms: conditions — Gender Dysphoria; Transsexualism | interventions — testosterone 17 beta-cypionate; Estradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transmen: Subjects starting testosterone therapy as part of standard of care for gender incongruence
  Interventions: Drug: testosterone cypionate
- transwomen: Subjects starting estradiol therapy as part of standard of care for gender incongruence
  Interventions: Drug: Estradiol Valerate

INTERVENTIONS:
Drug: testosterone cypionate — intramuscular injection every 2 weeks. Dose will be titrated based on blood levels
  Groups: Transmen
Drug: Estradiol Valerate — intramuscular injection every week. Dose will be titrated based on blood levels
  Groups: transwomen

SUMMARY:
The purpose of this research is to find out if hormone therapy in transgender subjects' changes hormone receptors in blood, muscle and fat; fat production; muscle production; and inflammation processes.

DETAILED DESCRIPTION:
Throughout recorded history, some men and women have experienced emotional distress at being physically "trapped" in wrong gender. Gender incongruence refers to the state where one's internal sense of gender differs from the gender assigned at birth. Advances in psychology and in our understanding of human sexuality have permitted the recognition of gender incongruence (also called transgender) as a biological phenomenon. The acceptance by the society has led to an expansion of health care services available to these individuals for supportive treatment. Gender affirming hormone therapy, usually provided by endocrinologists, is pivotal for the transition of these individuals into their desired gender. This therapy typically consists of testosterone or estrogen (male and female sex hormones) to transition into transmen or transwomen, respectively. The hormone treatment results in a "second puberty", wherein biological men receiving estrogen gain fat around hips and thighs, lose muscle and develop breasts. Biological women receiving testosterone lose fat, gain muscle, stop having menses and develop a deeper voice. However, our knowledge of the mechanisms of these hormones at the tissue level in transgender population is lacking. In this study, we plan to evaluate

1. hormone receptors that carry out the action of sex hormones in fat tissue and mononuclear cells (a type of immune cell in blood) following gender affirming therapy.
2. the mechanism that lead to growth or suppression of fat mass or lean mass
3. effect on inflammation (a cardiovascular risk marker) The hormone treatment of gender incongruence is a relatively untested therapy. The treatment is based on extrapolations and assumptions from hormone treatment in hypogonadal (hormone deficient) in cis-gender (same gender, no incongruence) individuals. We expect that our mechanistic studies will initiate an understanding into the actions of transgender therapy at the cellular level.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gender incongruence by a mental health professional and willing to start gender affirming therapy

Exclusion Criteria:

* Used hormone therapy in last 6 months,
* Pregnancy,
* Planning to have biological children in the next one year,
* HIV Additional exclusion criteria for transmen: 1) hematocrit >50% for transmen, 2) transmen with allergy to cottonseed oil (component of intramuscular testosterone injection), 3) uncompensated heart failure, 4) renal failure Additional exclusion criteria for transwomen: 1) allergy to castor oil (component of intramuscular estradiol injection), 2) Known or suspected estrogen-dependent neoplasia, 3) Active deep vein thrombosis, pulmonary embolism or a history of these conditions, 4) Active or recent (e.g., within the past year) arterial thromboembolic disease (e.g., stroke, myocardial infarction), 5) Liver enzymes (AST or ALT) >3 times the upper limit of normal, 6) Known or suspected pregnancy

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Gender Based: Yes — 2 groups based on gender identity: transowmen and transmen
Study Population: We plan to conduct a prospective, open label study in individuals initiating gender affirming therapy for gender incongruence. We will recruit 20 transmen and 20 transwomen in this study.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Androgen receptor | 6 months
  change in Androgen receptor expression in subcutaneous adipose tissue in transmen

SECONDARY OUTCOMES:
Estrogen receptor and aromatase | 6 months
  Expression and protein content of estrogen receptor alpha and aromatase in muscle and fat of transmen and transwomen
inflammation | 6 months
  expression of inflammatory mediators in fat tissue and circulating levels in serum
autophagy | 6 months
  Assessment of autophagic flux in fat and muscle biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Dhindsa, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis Univeristy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No